CLINICAL TRIAL: NCT06875128
Title: An Open-label, Randomized, Multi-Center Study to Evaluate the Efficacy and Safety of Induction Treatment With Melphalan/HDS Followed by Consolidation Treatment With Eribulin or Vinorelbine or Capecitabine Versus Eribulin or Vinorelbine or Capecitabine Alone in Patients With Metastatic Breast Cancer With Liver Dominant Disease
Brief Title: Evaluation of the Safety and Efficacy of Treatment w/High Dose Melphalan Given Directly Into the Liver Followed by Treatment w/Approved Cancer Treatment or Approved Cancer Treatment Alone in Patients w/ Metastatic Breast Cancer w/Liver Dominant Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Delcath Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHP-MBC-202
Record Dates: First submitted 2025-03-06; First posted 2025-03-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Breast Cancer in the Liver
Keywords: melphalan; melphalan/HDS; melphalan/hepatic delivery system; eribulin; vinorelbine; capecitabine; metastatic breast cancer; MBC; liver dominant disease; metastatic breast cancer in the liver; hepatic delivery system; PHP; HER2-negative breast cancer; HER-2 negative; Hormone Receptor-Positive disease
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Vinorelbine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melphalan/HDS followed by Physician's choice of SOC (eribulin, vinorelbine, or capecitabine) (Experimental): Melphalan/HDS is given as an infusion of Melphalan into the hepatic artery under general anesthesia. This treatment is administered then followed by Physician's choice of SOC (eribulin, vinorelbine, or capecitabine) then repeated for a second cycle of Melphanlan/HDS followed by Physician's choice of SOC.
  Interventions: Drug: Melphalan/HDS followed by Physician's choice of SOC (eribulin, vinorelbine, or capecitabine)
- Physician's choice of SOC (eribulin, vinorelbine, or capecitabine) Alone (Active Comparator): Physician's choice of SOC (eribulin, vinorelbine, or capecitabine)
  Interventions: Drug: Physician's choice of SOC (eribulin, vinorelbine, or capecitabine)

INTERVENTIONS:
Drug: Melphalan/HDS followed by Physician's choice of SOC (eribulin, vinorelbine, or capecitabine) — Melphalan/HDS followed by Physician's choice of SOC (eribulin, vinorelbine, or capecitabine)
  Arms: Melphalan/HDS followed by Physician's choice of SOC (eribulin, vinorelbine, or capecitabine)
Drug: Physician's choice of SOC (eribulin, vinorelbine, or capecitabine) — Physician's choice of SOC (eribulin, vinorelbine, or capecitabine)
  Arms: Physician's choice of SOC (eribulin, vinorelbine, or capecitabine) Alone

SUMMARY:
The goal of this clinical trial is to learn if using a liver-directed therapy with high dose chemotherapy followed by approved cancer treatment to treat patients with breast cancer that has spread to the liver is safe and tolerable. The clinical trial will also learn if the liver-directed therapy with high dose chemotherapy works on the disease in the liver. Investigators will compare the use of the liver-directed therapy with high dose chemotherapy followed by approved cancer treatment or approved cancer treatment alone.

Participants will:

* Undergo up to two cycles of liver-directed therapy with high dose chemotherapy procedures followed by approved cancer treatment or take approved cancer treatment alone
* Visit clinic at least every two weeks for checkups and tests
* Complete scans approximately every 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of MBC.
* Patients with HER2-negative (IHC 0 or 1+ or 2+ and ISH non-amplified) MBC (including triple negative disease).
* Patient with Hormone Receptor-Positive disease has progressed on or intolerant of prior endocrine therapy and CDK 4/6 inhibitors.
* Disease progression after TOPO-1 isomerase inhibitor payload ADC, such as sacituzumab govitecan and/or trastuzumab deruxtecan. Patients not eligible or suitable for ADCs can be considered for this study. NOTE: In jurisdictions where those ADCs are not available as standard of care, patients will be eligible after prior treatment or intolerable toxicity on two standard chemotherapy regimens for the appropriate disease subtype.
* Patient with HER2-negative breast cancer suitable for single agent chemotherapy as per judgement of treating investigator.
* Patient is a suitable candidate for treatment with one of the following: eribulin, vinorelbine, or capecitabine as per judgement of treating investigator.
* Patient has liver dominant metastatic disease. Liver-dominant is defined as the majority of total tumor burden is located in the liver, and/or the life-threatening component of the disease is located in the liver.
* MBC metastases must involve ≤ 50% of the liver parenchyma.
* If there is evidence of extrahepatic metastatic disease, it is limited, and the life-threatening component of disease is in the liver. Extrahepatic disease is restricted to lesions in the breast, lung, other visceral organs, lymph nodes and skin.
* Disease in the liver must be measurable (per RECIST v1.1 guidelines) by computed tomography (CT) and/or magnetic resonance imaging (MRI).
* Patient weighs ≥ 35 kg
* Scans used to determine eligibility (CT scan of the chest/abdomen/pelvis and MRI of the liver) must be performed within 28 days prior to randomization.
* Patient has an ECOG PS of 0-1.

Exclusion Criteria:

* Prior chemoembolization or radioembolization to the liver or prior hepatic arterial infusion therapy.
* Evidence of clinically significant portal hypertension by history, endoscopy, or radiologic studies (large abdominal varices, prior history of varices by endoscopy).
* New York Heart Association functional classification II, III or IV or active cardiac condition(s), including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), worsening or new-onset congestive heart failure, significant arrhythmias, or severe valvular disease that create(s) undue risks of undergoing general anesthesia.
* History or evidence of clinically significant pulmonary disease that precludes the use of general anesthesia.
* History of bleeding disorders, presence of brain metastases or other intracranial abnormalities that would put them at risk for bleeding with anti-coagulation.
* Known varices at risk of bleeding, including medium or large esophageal or gastric varices, active peptic ulcer, or history of recent hemoptysis.
* An active second malignancy or has a history of recent definitively treated invasive cancer within 2 years prior to enrolment. Exceptions are optimally treated and controlled basal cell carcinoma, other skin cancers, thyroid cancer.
* Symptoms and signs indicating clinically significant progression of disease including cord compression, increasing pain symptoms, increasing oxygen requirements, impending pathological fracture, compressive lymphadenopathy, or symptomatic pleural effusion.
* Pregnant or breastfeeding.
* WOCBP (i.e., fertile meaning not permanently sterilized and having had a menstrual period within the past 12 months) who is unable to undergo hormonal suppression to avoid menstruation during treatment.
* Patient requires chronic use of immunosuppressive drugs. NOTE: Oral prednisolone ≤ 10 mg/day or equivalent is allowed.
* Unable to be temporarily removed from chronic anti-coagulation therapy.
* Active bacterial infections with systemic manifestations (malaise, fever, leucocytosis).
* An active infection, including Hepatitis B and Hepatitis C infection. NOTE: Patients with anti-hepatitis B core antibody (HBc) positive, or hepatitis B surface antigen (HBsAg) but DNA negative are allowed exception(s).
* Known severe allergic reaction to iodine contrast that cannot be controlled by premedication with antihistamines and steroids.
* History of or known hypersensitivity to melphalan or the components of the Melphalan/HDS system.
* Known latex allergy.
* History of known hypersensitivity to heparin or the presence of heparin-induced thrombocytopenia.
* Uncontrolled endocrine disorder including diabetes mellitus, hypothyroidism, or hyperthyroidism.
* Received anti-cancer therapy including radiotherapy or investigational agent for any indication ≤ 30 days prior to randomization.
* Patients should have recovered to Grade 1 or less for AEs related to prior treatment unless deemed clinically not significant, such as lymphopenia, anemia, or grade 2 neuropathy due to prior taxane treatment.

NOTE: Certain side effects that are unlikely to develop into serious or life-threatening events (e.g., alopecia) are allowed at ≥ Grade 1.

* < 28 days after surgery and surgical wound is not fully healed.
* Currently under treatment for cancer other than MBC or is not deemed to be cancer free.
* Not eligible to receive either eribulin or vinorelbine or capecitabine.
* Albumin level < 3.0 g/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
hPFS | assessed through study completion, an average of 2 years
  Hepatic Progression Free Survival

SECONDARY OUTCOMES:
PFS | assessed through study completion, an average of 2 years
  Progression Free Survival
ORR | Baseline through completion of treatment, assessed through study completion, an average of 2 years
  Overall Response Rate complete response [CR] + partial response [PR]
hORR | assessed through study completion, an average of 2 years
  Hepatic Overall Response Rate
DOR | assessed through study completion, an average of 2 years
  Duration of Response
hDOR | assessed through study completion, an average of 2 years
  Hepatic duration of response
DCR | assessed through study completion, an average of 2 years
  Disease control rate
hDCR | assessed through study completion, an average of 2 years
  Hepatic disease control rate
OS | assessed through study completion, an average of 2 years
  Overall Survival

OTHER OUTCOMES:
Safety and Tolerability | assessed through study completion, an average of 2 years
  Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)
Pharmacokinetic Endpoint | assessed through study completion, an average of 2 years
  Local and systemic exposure of melphalan administered by the HDS

IPD SHARING:
Plan to Share IPD: No
Delcath does not currently have a plan to share IPD.